CLINICAL TRIAL: NCT04248972
Title: Short- and Long-term Effects of Photobiomodulation on Pain, Functionality, Tissue Quality, Central Sensitisation and Psychological Factors in a Population Suffering From Fibromyalgia: Protocol for a Triple-blinded Randomized Clinical Trial.
Brief Title: Effects of Photobiomodulation in a Population Suffering From Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, SANTIAGO NAVARRO LEDESMA, UNIVERSITY PROFESSOR, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBMFM
Record Dates: First submitted 2020-01-18; First posted 2020-01-30 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Fibromyalgia; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): A treatment with whole body red light therapy (NovoTHOR®) will be carried out
  Interventions: Device: PBM
- PLACEBO INTERVENTION (Placebo Comparator): A placebo whole body red light will be carried out
  Interventions: Other: PLACEBO PBM

INTERVENTIONS:
Device: PBM — A whole body red light therapy (NovoTHOR®) will be carried out during 20 minutes
  Arms: Intervention
Other: PLACEBO PBM — A placebo whole body red light will be carried out during 20 minutes
  Arms: PLACEBO INTERVENTION

SUMMARY:
The development of an integral and global treatment to improve the quality of life in those with fibromyalgia syndrome (FMS) is challenging, thus a whole body Photobiomodulation (PBM) therapy program is proposed as an effective option.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled clinical trial. Participants will be recruited in a private care practice and randomized to receive either a whole body Photobiomodulation (PBM) therapy program or placebo. Primary outcomes will be pain (Numeric Pain Rating Scale; Widespread Pain Index; Symptom Severity Score), functionality (Fibromyalgia Impact Questionnaire; The Leisure Time Physical Activity Instrument), quality of soft tissue (elastography) and central sensitisation (pain pressure threshold and the Autonomic Symptom Profile). Secondary outcomes will be psychological factors (Pain Catastrophising scale, Tampa Scale, Self-Efficacy questionnaire). Assessments will be at baseline, after treatment 6, immediately following the last treatment (4 weeks), and then 2 weeks and at 3 monthly follow up intervals to 6 months after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed from FM presenting generalized pain in at least four or five regions.
* Present symptoms for at least 3 months at similar levels.

Exclusion Criteria:

- Inflammatory, neurological, or orthopedic disease which can alter balance, hearing, and vision, and cognitive impairment in terms of the ability to answer questions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline perceived pain at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Visual Analogue Scale (VAS) is used by the patient to quantify the pain from 0 (without any pain) to 10 (the worst pain)
Change from baseline Leisure Time Physical Activity Instrument (LTPAI) at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  The Leisure Time Physical Activity Instrument (LTPAI), used to measure the physical activity. This has four components, each with three levels of activity: light, medium, and vigorous. Scores indicate the number of hours which these activity levels had been carried out each week in the last four weeks summing as the total number of hours of physical activity
Change from baseline Widespread Pain Index (WPI) at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Widespread Pain Index (WPI) is a questionnaire which shows appropriate distribution and a sufficient number of body quadrants and axial skeleton pain representation. It is part of the FMS diagnosis.
Change from baseline Symptom Severity Score (SSS) at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Symptom Severity Score (SSS) is a questionnaire whichispart of the FMS diagnosis
Change from baseline Impact Questionnaire (FIQR) at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  The revised Fibromyalgia Impact Questionnaire (FIQR), a self-administered questionnaire comprising 21 individual questions, with a rating scale of 0-10. The questions compose three different domains: function, overall impact and symptoms score (range 0-30, 0-20 and 0-50, respectively). The FIQR total score ranges from 0 to 100, with a higher score indicating a greater impact of the condition on the person'slife.
Change from baseline Pain pressure threshold in neck and upper limb at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Tender points will be assessed using a standard pressure algometer (FPK 20; Wagner Instruments, Greenwich, CT, USA.): occiput at the suboccipital muscle insertions, low cervical at the anterior aspects of the intertransverse spaces at C5-C7, trapezius at the midpoint of the upper border, supraspinatus at origins, above the scapula spine near the medial border, paraspinous 3 cm lateral to the midline at the level of the mid-scapula, second rib at the second costochondral junctions, just lateral to the junctions on the upper surfaces, lateral pectoral at the level of the fourth rib at the anterior axillary line, lateral epicondylee 2 cm distal to the epicondyles and medial epicondyle at the epicondyles.
Change from baseline Pain pressure threshold in lower limb at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Tender points will be assessed using a standard pressure algometer (FPK 20; Wagner Instruments, Greenwich, CT, USA.): gluteal at the upper outer quadrants of buttocks in anterior fold of muscle, greater trochanter just posterior to the trochanteric prominence, and knees at the medial fat pad proximal to the joint line, forearm at the distal dorsal third of the forearm, thumbnail, and midfoot at the midpoint of the dorsal third metatarsal.
Change from autonomic nervous system activity at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  The Autonomic Symptom Profile (ASP) is a validated self-report questionnaire that comprehensively assesses autonomic symptoms across 11 subscales and yields a composite autonomic symptom score, where higher scores mean a better outcome and lower scores mean a worst outcome. Autonomic nervous system activity provides quantitative information regarding cardiac autonomic tone.
Change from elastography at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Quantified elastography in tender points. Changes in the status of myofascial trigger-points can be demonstrated with an objective and reproducible USE measure

SECONDARY OUTCOMES:
Change from baseline Pain catastrophizing Scale (PCS) at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Assessment of the mechanisms by which catastrophizing impacts on pain experience. Higher scores mean a better outcome and lower scores mean a worst outcome.
Change from baseline kinesiophobia at 6 months | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  Assessment of the fear of movement through the validated Tampa-Scale questionnaire.
  Higher scores mean a better outcome and lower scores mean a worst outcome.
Change from baseline self efficacy questionnaire at 6 month | time (t) 1(prior to treatment), t2 (immediately after treatment 6), t3 (3 immediately following the last treatment), t4 (2 weeks after completion of treatment), t5 ( 3 months after completion of treatment), t6 ( 6 months after completion of treatment)
  The Self Efficacy Questionnaire assesses personal confidence to carry out an activity with the aim of successfully achieving a desired outcome.
  Higher scores mean a better outcome and lower scores mean a worst outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain

REFERENCES:
- [Derived] Navarro-Ledesma S, Gonzalez-Munoz A, Carroll J, Burton P. Short- and long-term effects of whole-body photobiomodulation on pain, functionality, tissue quality, central sensitisation and psychological factors in a population suffering from fibromyalgia: protocol for a triple-blinded randomised clinical trial. Ther Adv Chronic Dis. 2022 Feb 21;13:20406223221078095. doi: 10.1177/20406223221078095. eCollection 2022. PMID 35222905